CLINICAL TRIAL: NCT07180264
Title: Trastuzumab Deruxtecan in Patients With Advanced Breast Cancer: a Real-world Study
Brief Title: Trastuzumab Deruxtecan in Advanced Breast Cancer
Status: Recruiting | Type: Observational
Sponsor: Wenjin Yin (Other)
Responsible Party: Sponsor-Investigator, Wenjin Yin, Deputy Chief of Breast Surgery Department, RenJi Hospital
Organization: RenJi Hospital (Other)
Other Study IDs: LY2025-137-B
Record Dates: First submitted 2025-09-11; First posted 2025-09-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Advanced Breast Cancer
MeSH Terms: interventions — trastuzumab deruxtecan

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Trastuzumab deruxtecan: Trastuzumab deruxtecan, recommended dose 5.4mg/kg, every 21 days
  Interventions: Drug: Trastuzumab deruxtecan

INTERVENTIONS:
Drug: Trastuzumab deruxtecan — Trastuzumab deruxtecan is a combination of the targeted cancer drug trastuzumab (also known as Herceptin) and a chemotherapy drug called deruxtecan or DXd.

SUMMARY:
To evaluate the efficacy and safety of trastuzumab deruxtecan in advanced breast cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 and older
* Breast cancer patients meeting current guideline recommendations and planning to receive trastuzumab deruxtecan
* ECOG 0-1

Exclusion Criteria:

* During pregnancy and lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Breast cancer patients meeting current guideline recommendations and planning to receive trastuzumab deruxtecan
Sampling Method: Non-Probability Sample
Enrollment: 118 (Estimated)
Dates: Start 2025-08-28 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | From the date of starting Disitamab vedotin to the date of first documentation of progression or death (up to approximately 1 years)
  The time from the date of starting trastuzumab deruxtecan to the date of disease progression as per RECIST version 1.1 or death from any cause, whichever occurs first.

SECONDARY OUTCOMES:
Adverse events | From the date of starting trastuzumab deruxtecan to the end of the treatment (up to approximately 1 year)
  Adverse events during trastuzumab deruxtecan will be assessed according to the NCI CTCAE v5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Wenjin Yin, M.D., Principal Investigator — Renji Hospital,School of Medicine, Shanghai Jiaotong University
Locations (1):
- Renji Hospital, School of Medicine, Shanghai Jiaotong University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No